CLINICAL TRIAL: NCT04247841
Title: Remembering Risk: Using Visual Risk Display of MINS to Obtain Informed Consent to Undergo Elective Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. Michael McMullen (Other)
Responsible Party: Sponsor-Investigator, Dr. Michael McMullen, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TRAQ #: 6028012
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Risk
Keywords: Risk; Preoperative Assessment; Myocardial Injury; Perioperative Medicine; Personalized Medicine; Communication
MeSH Terms: conditions — Communication | interventions — Audiovisual Aids

STUDY DESIGN:
Intervention Model Description: During Phase 1 we will be completing data collection on a prospective cohort of patients attending Presurgical Screening (PSS) Clinic in preparation for elective total joint arthroplasty of the hip or knee.
  During the Phase 2 we will utilize a randomized approach to generate 2 groups of patients who will have their preoperative risk discussion guided by the use of a structured script or have the risk discussion guided by the use of a structured script and the display of a visual aid outlining the risk of myocardial injury
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be masked to the primary purpose of the study during their preoperative consultation. Upon receiving and completing the survey responses they will be asked to recall their individualized risk of myocardial injury and provide feedback on the risk discussion they had with the anesthesiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase I: Current Practice (No Intervention): This represents the first phase of the study in which a prospective cohort of patients will complete the survey to define baseline rates of recall of perioperative risk and level of patient satisfaction with risk discussion
- Phase II Visual Aid & Scripted Risk Discussion (Experimental): This will involve a group of patients randomized to receive their perioperative risk discussion supplemented with the use of a visual aid in addition to a scripted discussion of their personalized perioperative risk of myocardial injury (MINS) during their consultation with an anesthesiologist in the PSS clinic.
  Interventions: Other: Visual Aid; Other: Scripted Risk Discussion
- Phase II Scripted Risk Discussion (Active Comparator): This will involve a group of patients randomized to receive a scripted discussion of their personalized perioperative risk of myocardial injury (MINS) during their consultation with an anesthesiologist in the PSS clinic.
  Interventions: Other: Scripted Risk Discussion

INTERVENTIONS:
Other: Visual Aid — The visual aid will include a graphic display of 100 individuals with number of individuals anticipated to suffer a myocardial injury highlighted by being filled in in red. There will also be a textual discription stating the anticipated risk. For example in a patient with an rCRI score = 2 the text will state 10 out of 100 patients will have a myocardial injury (MINS) and 90 out of 100 patients will have no myocardial injury and 10 of the patients will be shaded red on the visual aid. The patients in this intervention will also received the scripted discussion of perioperative risk of MINS.
  Arms: Phase II Visual Aid & Scripted Risk Discussion
Other: Scripted Risk Discussion — The patients seen in PSS will have a standardized discussion of perioperative risk of myocardial injury read to them by the anesthesiologist in the PSS clinic.
  Arms: Phase II Scripted Risk Discussion; Phase II Visual Aid & Scripted Risk Discussion

SUMMARY:
Disclosure of anticipated risks to individuals considering undergoing an operative procedure is an important aspect of informed consent process. Recent Canadian Guidelines have highlighted the importance of perioperative risk discussion within the context of preoperative assessment but there is little prior research into potential interventions to optimize the communication of risks. Myocaridal injury (MINS) is the most common complication and this study is focused on determining the effectiveness of current communication strategies in our presurgical consultations and to quantifying the impact of introducing a visual aid and scripted risk discussions has on patients ability to recall their individualized perioperative risk of myocardial injury.

DETAILED DESCRIPTION:
Informed consent is an important aspect of the patient-physician relationship. Prior to agreeing to undergo treatment patients must have risks and benefits disclosed to a "reasonable patient" standard.1 The 2016 Canadian Cardiovascular Society Guidelines on Perioperative Cardiac Risk Assessment strongly recommend the communication of perioperative cardiac risk to patients.2 Myocardial injury is the most common post-operative complications and has significant impact on patient outcomes including survival.2. However, very few studies have examined the communication of risk to patients, particularly when communicating perioperative cardiac risk.

The aim of this study is a 2-stage research project to address current practice in perioperative risk communication and examine opportunity to improve communication and patient education.

Phase One is structured to assess the current practices with respect to cardiac risk discussion at our academic center. During this initial phase, a survey will be offered after the PSS consultation to patients > 45 years old, seen in consult prior to elective orthopedic surgery requiring an overnight admission to KHSC. The survey will assess current risk discussion practices, patient satisfaction with cardiac risk discussion, ability to recall cardiac risk, importance of cardiac risk disclosure, and seek general feedback from participants.

Phase Two of this study is structured to assess the effectiveness of incorporating the use of structured, scripted risk discussion with and without the use of a visual aid. The patients will complete the survey instrument immediately after their PSS consultation to assess patient satisfaction with cardiac risk discussion, recall of risk, importance of cardiac risk discussion from the patients' perspective, and general feedback will be sought regarding perioperative education.

A subset of consenting patients during both Phase I and II will be followed-up post operatively (within 48h) to assess recall of preoperative cardiac risk discussion.

Our study group hypothesizes that the use of visual representation of perioperative risk of Myocardial Injury after Non-Cardiac Surgery during the pre-anesthetic assessment will improve the patients' satisfaction with the cardiac risk discussion and their understanding and retention of the risk in the post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients 45 years of age or older who are seen in Presurgical Screening Clinic by an anesthesiologist prior to elective hip or knee arthroplasty at Kingston Health Sciences Centre.

Exclusion Criteria:

* Unable to provide consent due to communication/language barrier
* Prior enrollment in this study
* No planned admission to hospital ( Same - Day joint arthroplasty)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Immediate Recall of Perioperative Risk of Myocardial Injury (MINS) | Within 60 minutes of completing consultation with anesthesiologist in PSS clinic
  This will be calculated as the patients who can state their risk estimate within the 95% CI for the risk estimate given their rCRI score (as outlined in the 2016 CCS Guidelines) when completing the survey.

SECONDARY OUTCOMES:
Postoperative Recall of Perioperative Risk of Myocardial Injury (MINS) | Within 48 hours of undergoing their elective joint arthroplasty
  This will be calculated as the patients who can state their risk estimate within the 95% CI for the risk estimate given their rCRI score (as outlined in the 2016 CCS Guidelines) when completing the survey.
Demographics and Immediate Recall of Perioperative Risk of Myocardial Injury | Within 60 min of completing preoperative consultation
  We will compare the impact sex, age and level of education have on the percentage of patients able to recall their risk estimate within the 95% CI outlined in CCS guidelines
Correlation between subjective rating of individual risk and numeric risk estimate | Within 60 min completing preoperative consultation
  Patients subjective responses to their level of risk (minimal, low, moderate, high, very high) will be compared with their numeric risk estimate ( rate / 100 persons)
Satisfaction with Risk Discussion | Within 60 min completing preoperative consultation
  Subjects will be asked to rate their level of satisfaction with the preoperative risk discussion on a 5 point Likehert Scale and the difference between 3 arms will be examined
Recommendation of Use of Risk Discussion Tool in Future | Within 60 min completing preoperative consultation
  Patients will be asked to rate their likelihood (0-10) to use a similar format of risk discussion to family or friends coming for surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McMullen, MD, Principal Investigator — Department of Anesthesiology and Perioperative Medicine, Queen's Univerisity
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No